CLINICAL TRIAL: NCT05318703
Title: Virtual Exercise Intervention for Older Adults With MCI
Brief Title: Virtual Exercise For Older Adults With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AG059546-02S1
Record Dates: First submitted 2022-03-23; First posted 2022-04-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Mild Cognitive Impairment
Keywords: tai chi, ehealth, older adults, cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitively enhanced tai ji quan (Experimental): Participants receive a cognitively enhanced tai ji quan exercise intervention for 16 weeks.
  Interventions: Behavioral: tai ji quan
- stretching exercise (Active Comparator): Participants receive a stretching exercise intervention for 16 weeks.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: tai ji quan — cognitively enhanced tai ji quan exercise
  Arms: cognitively enhanced tai ji quan
Behavioral: Stretching — Stretching exercise
  Arms: stretching exercise

SUMMARY:
This project is designed to develop and evaluate an Internet-based exercise intervention (tai ji quan Moving to Improve Brain Health) using real-time videoconferencing for older adults with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The project has three major goals: (a) transforming an in-person tai ji quan brain health intervention protocol into an online (virtual) class protocol and evaluating its feasibility of implementation in older adults with MCI, (b) developing and evaluating online assessment and data ascertainment procedures that encompass cognitive and physical performance measures, and (c) conducting a randomized controlled trial comparing the effectiveness of this new online intervention protocol with a conventional stretching exercise group in older adults with MCI.

ELIGIBILITY:
Inclusion criteria:

* Self-report a change or decline in memory (corroborated by an informant)
* Record a score of ≤0.5 on the Clinical Dementia Rating (CDR) scale (with information derived from both the participant and an informant)
* Show no major impairment in cognitive function as indexed by a score of ≥24 on the Mini Mental State Evaluation (MMSE).

Exclusion criteria:

* Have participated in a rigorous and structured physical activity or exercise program (including Tai Ji Quan) in the past 6 months,
* Show major signs of depression as indicated by a score of ≥5 on the Geriatric Depression Scale
* Have major medical or physical conditions that preclude exercise, as determined by their healthcare practitioner
* Being unable to follow the consent process or sign the study consent form.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
(a) Total number of intervention sessions taught by instructors over the course of study (recorded by a class check sheet) and (b) total number of classes attended by participants over the course of intervention as recorded by class attendance sheet | 16 weeks
  assess the extent to which interventionists successfully implement the prespecified exercise training protocol.
number of dropouts from the intervention and study as assessed by a study recording sheet | 16 weeks
  assess intervention dropout rate and retention rate
Number of participants expressing intervention program satisfaction as assessed by a self-report survey | 16 weeks
  assess the program acceptability among tai ji quan participants
Change in global cognitive function assessed by Montreal Cognitive Assessment | baseline, 16 weeks
  assess change from baseline cognitive function at 16 weeks
Change in attention and working memory as assessed by Digit Span - forward and backward | baseline, 16 weeks
  assess change from baseline in attention and working memory at 16 weeks
Change in dual-task cost as assessed by Timed Up and Go with a cognitive task | baseline, 16 weeks
  assess change from baseline in the ability to stand up from a chair, walk, and sit down while performing an arithmetic task at 16 weeks
Change in executive function as assessed by Trail Making B | baseline, 16 weeks
  assess change from baseline executive function at 16 weeks
Change in executive function as assessed by Category Fluency for Animals | baseline, 16 weeks
  assess change from baseline executive function at 16 weeks
Change in cognitive functioning assessed by Everyday Cognition | baseline, 16 weeks
  assess change from baseline cognitive functioning at 16 weeks
Change in physical performance as measured by Timed Up and Go test | baseline, 16 weeks
  assess change from baseline in the ability to stand up from a chair, walk, and sit down at 16 weeks
change in leg strength as assessed by 30-second chair stand test | baseline, 16 weeks
  assess change from baseline in leg strength at 16 weeks
Change in balance using a 4-stage balance test | baseline, 16 weeks
  assess change from baseline in balance at 16 weeks

SECONDARY OUTCOMES:
Change in depression as assessed by Geriatric Depression scale | baseline, 16 weeks
  assess change from baseline in the level of depression at 16 weeks
Change in physical activity as assessed by International Physical Activity Questionnaire | baseline, 16 weeks
  assess change from baseline in physical activity at 16 weeks
Change in quality of life as assessed by EuroQol (EQ-5D-3L) | baseline, 16 weeks
  assess change from baseline in quality of life at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fuzhong Li, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol
Time Frame: 12 months after the completion of the study.
Access Criteria: The de-identified data that support the findings of this study are available from the corresponding author upon reasonable request. Restrictions may apply to preserve participant confidentiality.